CLINICAL TRIAL: NCT06946368
Title: A Single-Center, Randomized, Pilot Study to Assess the Clinical Effectiveness of EXPAREL as an Intra-articular Posteromedial Surgeon Administered (IPSA) Block in Subjects Undergoing Primary Unilateral Total Knee Arthroplasty
Brief Title: Effectiveness of Exparel Anesthetic Administered by the Surgeon During Knee Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-033
Record Dates: First submitted 2025-04-16; First posted 2025-04-27 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Total Knee Arthroplasty
Keywords: Exparel; Primary Unilateral Total Knee Arthroplasty; IPSA block

STUDY DESIGN:
Intervention Model Description: This is a randomized pilot study. The study will enroll 60 total subjects 1:1:1 to receive treatment on the day of surgery.
  The randomization code will be computer-generated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Patients in this group will receive IPSA block and Local Infiltration Analgesia (LIA).
  Interventions: Procedure: Intra-articular Posteromedial Surgeon Administered (IPSA) Block of EXPAREL
- Group 2-Control (Standard of Care) (Active Comparator): Patients in this group will receive Adductor Canal Block (ACB) and Local Infiltration Analgesia (LIA).
  Interventions: Procedure: Adductor Canal Block (ACB) and Local Local Infiltration Analgesia of EXPAREL
- Group 3 (Experimental): Patients in this group will receive Local Infiltration Analgesia (LIA).
  Interventions: Procedure: Local Infiltration Analgesia (LIA) of EXPAREL

INTERVENTIONS:
Procedure: Intra-articular Posteromedial Surgeon Administered (IPSA) Block of EXPAREL — Patients in this group will receive IPSA block and Local Infiltration Analgesia (LIA).
  IPSA block is a pain numbing medication given by surgeon and injected inside the back and inner side of the knee joint. Local Infiltration Analgesia is a pain numbing medication injection given by the surgeon around the surgical knee area. The medications used in the procedure will be EXPAREL, and Bupivacaine HCL.
  Arms: Group 1
Procedure: Adductor Canal Block (ACB) and Local Local Infiltration Analgesia of EXPAREL — ACB is a pain numbing injection given by anesthesiologist near the adductor canal, a passage in the mid-thigh that contains nerves connecting the knee region. Local Infiltration Analgesia is a pain numbing medication injection given by the surgeon around the surgical knee area. The medications used in the procedure will be EXPAREL, and Bupivacaine HCL.
  Arms: Group 2-Control (Standard of Care)
Procedure: Local Infiltration Analgesia (LIA) of EXPAREL — Local Infiltration Analgesia is a pain numbing medication injection given by the surgeon around the surgical knee area. The medications used in the procedure will be EXPAREL, and Bupivacaine HCL.
  Arms: Group 3

SUMMARY:
Intra-articular Posteromedial Surgeon Administered (IPSA) Block in this study describes a new type of medical procedure where a surgeon provides anesthetic medication directly into a specific area inside a knee joint to numb the pain during knee surgery. Intra-articular refers to inside of knee joint, posteromedial refers to the back and inner side of a knee joint, and surgeon administered means a surgeon is performing the procedure.

Patients You will be randomly assigned to one of these three treatment groups:

Group 1:

Patients in this group will receive IPSA block and Local Infiltration Analgesia (LIA).

IPSA block is a pain numbing medication given by surgeon and injected inside the back and inner side of the knee joint. Local Infiltration Analgesia is a pain numbing medication injection given by the surgeon around the surgical knee area. The medications used in the procedure will be EXPAREL, and Bupivacaine HCL.

Group 2 (Control):

Patients in this group will receive Adductor Canal Block (ACB) and Local Infiltration Analgesia (LIA). ACB is a pain numbing injection given by anesthesiologist near the adductor canal, a passage in the mid-thigh that contains nerves connecting the knee region. Local Infiltration Analgesia is a pain numbing medication injection given by the surgeon around the surgical knee area. The medications used in the procedure will be EXPAREL, and Bupivacaine HCL.

Group 3:

Patients in this group will receive Local Infiltration Analgesia (LIA). Local Infiltration Analgesia is a pain numbing medication injection given by the surgeon around the surgical knee area. The medications used in the procedure will be EXPAREL, and Bupivacaine HCL.

The study will evaluate;

* How effective the pain relief is after surgery.
* How much extra pain medication you need.
* Your satisfaction with pain management and recovery
* Any side effects.

DETAILED DESCRIPTION:
The study is a single-center, randomized, pilot study and will recruit up to 60 adult subjects undergoing unilateral total knee arthroplasty. Subjects will be randomized (1:1:1) to receive the treatments. The study participants will be followed for up to 90 days.

Information on analgesic use, pain, satisfaction with pain management will be obtained from patients. Participation begins when you sign the consent form. The treatment will begin on the day of the surgery. Follow up calls will be done 14 days and 90 days after surgery. Your involvement will last about 123 days.

Background and Rationale for the Study:

This study is being conducted to evaluate the clinical effectiveness of the Intra-articular Posteromedial Surgeon Administered (IPSA) block in subjects undergoing total knee arthroplasty (TKA). This study aims to demonstrate that a surgeon administered IPSA block can provide equivalent pain control to an anesthesiologist administered adductor canal block (ACB).

Method of Assigning Subjects to Treatment Randomization Scheme

Randomization Procedures Once a subject is identified as being qualified for the study in accordance with the eligibility criteria, the Investigator or designee will obtain a randomization assignment on the day of surgery. The subject will be considered randomized to the study once the study treatment is assigned.

Replacement of Subjects Subjects who withdraw from the study before the study treatment procedure may be replaced. Once a subject number is assigned, subject numbers will not be reused; subjects enrolled to replace those who withdraw will be assigned a unique subject number and randomized to treatment according to the procedures outlined above.

Subjects who are randomized but are withdrawn from the study before receiving the study drug may be replaced. Additionally, subjects may be replaced if insufficient and/or incomplete data are noted on safety or clinical outcomes.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation:

1. Subjects ages 18 or older at screening 2. Indicated to undergo primary unilateral total knee arthroplasty under spinal anesthesia 3. Primary indication for TKA is degenerative osteoarthritis of the knee 4. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3 (see Appendix 6) 5. Able to provide informed consent, adhere to the study schedule, and complete all study assessments 6. Body Mass Index (BMI) ≥18 and <40 kg/m2

-

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will not be eligible for participation in this study:

  1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine HCl, NSAIDs)
  2. Planned concurrent surgical procedure (e.g., bilateral TKA)
  3. Undergoing unicompartmental TKA or revision TKA
  4. Concurrent painful physical condition (e.g. arthritis, fibromyalgia, cancer) that may require analgesic treatment with NSAIDs or opioids in the post dosing period for pain that is not strictly related to the knee surgery and which, in the Investigator's opinion, may confound the post dosing assessments
  5. Inadequate sensory function below the knee as assessed by the Investigator
  6. History of contralateral TKA within 1 year
  7. Previous open knee surgery on the knee being considered for TKA. Prior arthroscopy is permitted
  8. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
  9. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
  10. Previous participation in an EXPAREL study
  11. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, could interfere with study assessments or compliance
  12. Currently pregnant, nursing, or planning to become pregnant during the study
  13. Clinically significant medical disease that, in the opinion of the Investigator, would make participation in a clinical study inappropriate. This includes diabetic neuropathy, coagulation or bleeding disorders, severe peripheral vascular disease, renal insufficiency, hepatic dysfunction or other conditions that would constitute a contraindication to participation in the study.
  14. Any use of marijuana [including Tetrahydrocannabinol (THC) and Cannabidiol (CBD)] within 30 days prior to randomization, or planned use during the course of the study
  15. Chronic opioid use (average ≥30 oral morphine equivalents/day) within 30 days prior to surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Questionnaires to assess the Pain levels of subjects enrolled in the study | 120 days
  Patients answer survey questionnaires about knee pain and general health. Pain levels will be taken regularly at 8, 24, 48 and 72 hours after surgery at the healthcare facility. Follow up questionnaire on pain levels will be done at 14 days and 90 days post-surgery. Patients share how satisfied they are with pain management at 72 hours, 14 days and 90 days after surgery.
  Subject's Reported Pain (Numeric Rating Scale) Pain intensity scores Subject will evaluate their pain in the operative knee using an 11-point Numeric Rating Scale (NRS), where 0=no pain and 10=worst possible pain.
Evaluate safety and any side effects | 120 days
  Record any (i.e., adverse events [AEs]) related to the EXPAREL IPSA block for the enrolled subjects.
Medication usage | 120 days
  Information about concomitant medication usage including opioids and analgesics
Subject Satisfaction Assessments | 120 days
  Subject Satisfaction Assessments (Likert Scale) Subject Satisfaction with Pain Management
  Overall satisfaction with your pain management. (Select one number only)
  1. Extremely dissatisfied
  2. Dissatisfied
  3. Neither satisfied nor dissatisfied
  4. Satisfied
  5. Extremely satisfied
Knee and general health survey | 120 days
  Questionnaires on knee health and general health. KOOS JR : Knee function will be assessed by the KOOS-JR questionnaire Forgotten Joint Score - 12: Joint Awareness questionnaires The Veterans RAND 12 Item Health Survey (VR-12): Health related quality of life will be assessed by the VR-12
Body Mass Index | 120 days
  weight and height measurements will be taken and calculated to report BMI in kg/m^2).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Deren, MD, Principal Investigator — Associate Staff Orthopaedic Surgery
Locations (1):
- Cleveland Clinic Lutheran Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Y, Huang Z, Ma W. Comparison of adductor canal block with local infiltration analgesia in primary total knee arthroplasty: A meta-analysis of randomized controlled trials. Int J Surg. 2019 Sep;69:89-97. doi: 10.1016/j.ijsu.2019.07.024. Epub 2019 Jul 30. PMID 31374265
- [Background] Piuzzi NS, Spitzer AI, Mussell J, Pasqualini I, Dysart S, Gonzales J, Mont MA, Lonner JH, Mihalko W. Validation of a Novel Landmark-guided Intra-articular Postero-medial Surgeon-administered Injection Technique. Arthroplast Today. 2025 Jan 25;31:101619. doi: 10.1016/j.artd.2025.101619. eCollection 2025 Feb. PMID 39927121